CLINICAL TRIAL: NCT01834222
Title: Post Marketing Surveillance To Observe Safety Of Prevenar 13 In Adults
Brief Title: Post Market Surveillance to Observe Safety of Prevenar13™ in Adults
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851143
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Korean adults aged 50 years and older who receive Prevenar13™ in a routine clinical setting
  Interventions: Biological: Non-intervention

INTERVENTIONS:
Biological: Non-intervention — Non-intervention

SUMMARY:
The purpose of this study is to assess safety profile of Prevenar 13™ when used among Korean adults in the routine clinical setting, as required for any new drug approved by Korea Food and Drug Administration (KFDA).

DETAILED DESCRIPTION:
non-randomization, non-probability sampling

ELIGIBILITY:
Inclusion Criteria:

Korean adults aged 18 years and older; provided the conditions pertaining to contraindications, warnings, precautions, and interactions stated in the local product document do not apply.

* Evidence of a personally signed and dated informed consent document indicating that the subject(or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

Subjects who are not indicated and/or contraindicated for the Prevenar13 usage will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean adults aged 18 years and older who receive Prevenar13™ in a routine clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- South Korea (25):
  - Chungnam National University Hospital (CNUH), Jung-gu, Daejeon
  - Bundang 21st Clinic, Seongnam-si, Gyeonggi-do
  - Lee soo yang Internal Medical Clinic, Guro-gu, Seoul
  - Hansarang Internal Medicine Hospital, Busan, South Korea
  - Shin Clinic Internal Medicine, Seoul, South Korea
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Samsung Happy Clinic, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Pusan National Univeristy Hospital, Daejeon
  - MiSo Medical, Daejeon
  - Sun's internal medicine, Daejeon
  - Techno Internal Medicine Clinic, Daejeon
  - Chuncheon Sacred Heart Hospital-Hallym University, Gangwon-do
  - Dr. Lee's Medical Clinic, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Suh Jeong Min Clinic, Gyeonggi-do
  - Bundang 21st Clinic, Gyeonggi-do
  - Light & Salt Internal Medicine, Gyeonggi-do
  - Seoul Samsung Medical Clinic, Seoul
  - Dr. Lee's Clinic of Internal Medicine, Seoul
  - Sung's Medical Clinic, Seoul
  - GF Internal Medicine, Seoul
  - Jong Koo Lee Heart Clinic, Seoul
  - Ulsan University Hospital, Ulsan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851143&StudyName=Post%20Marketing%20Surveillance%20To%20Observe%20Safety%20Of%20Prevenar%2013%20In%20Adults

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar 13: Participants received single dose of Prevenar 13 vaccine, 0.5 milliliter (mL) intramuscularly on Day 1. Participants were followed up to 28 days after last dose of study vaccination.
Period: Overall Study
Arm/Group | Prevenar 13
Started | 659
Treated | 658
Completed | 658
Not Completed | 1
Not completed — Not meet inclusion/exclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of Prevenar 13.
Groups:
- Prevenar 13: Participants received single dose of Prevenar 13 vaccine, 0.5 mL intramuscularly on Day 1. Participants were followed up to 28 days after last dose of study vaccination.
Arm/Group | Prevenar 13
Number analyzed (Participants) | 658
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.81 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337
  Male | 321

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose (up to Day 29) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AE.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of Prevenar 13.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 658
participants
  AEs | 140
  SAEs | 2

2. Primary Outcome: Duration of Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Duration of adverse event (in days) was defined as total time from onset of adverse event till the event was resolved during study.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of Prevenar 13.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prevenar 13
Number analyzed (Participants) | 658
days | 4.89 (7.22)

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AE was assessed on basis of severity as follows: a) mild: did not caused any significant problem to the participant; b) moderate: caused problem that did not interfere significantly with usual activities or the clinical status, other therapy needed due to AE; c) severe: caused problem that interfered significantly with usual activities or the clinical status.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of Prevenar 13.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 658
participants
  Mild | 127
  Moderate | 17
  Severe | 2

4. Primary Outcome: Number of Participants With Outcome in Response to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Outcome of an AE was assessed among participants based on their response to a question 'Is the adverse event still present?' as 'yes', 'unknown' or 'no (resolved)' during study.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety analysis set included all participants who received at least 1 dose of Prevenar 13. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 140
participants
  No (Resolved) | 132
  Yes | 3
  Unknown | 5

5. Primary Outcome: Number of Participants Who Discontinued Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline (Day 1) up to Day 29
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 140
participants | 0

6. Primary Outcome: Percentage of Adverse Events (AEs) With Their Causal Relationship to Study Drug
Description: Criteria: a)Certain: followed a reasonable time sequence from administration of drug; unexplained by other drugs, chemical substance or accompanying diseases;had clinically reasonable reaction on cessation of drug; had pharmacological or phenomenological reaction to re-administration of drug, b)Probable: followed a reasonable time sequence from administration of the drug; unexplained by other drugs;chemical substance or accompanying diseases; had clinically reasonable reaction on cessation of the drug, c)Possible:followed a reasonable time sequence from administration of drug; can also be explained by other drugs;chemical substance or accompanying diseases; lacks information or had unclear information on discontinuation of drug, d)Unlikely:not likely to had a reasonable causal relationship from administration of drug; seemed temporary; can also be reasonably explained by other drugs; chemical substances or latent diseases; conditional (need more data for true assessment),unaccessible.
Time Frame: Baseline (Day 1) up to Day 29
Population: as for outcome 4
Measure: Number; unit: percentage of adverse events
Arm/Group | Prevenar 13
Number analyzed (Participants) | 140
percentage of adverse events
  Certain | 47.60
  Probable | 24.04
  Possible | 20.67
  Unlikely | 7.69

ADVERSE EVENTS:
Description: The same event may appear as both AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experience both a serious and non-serious event during the study. Analysis was performed on safety analysis set.
Arm/Group | Prevenar 13
Serious Adverse Events (participants affected / at risk) | 2/658
Other Adverse Events (participants affected / at risk) | 139/658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=658)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
INFECTION VIRAL (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=658)
CELLULITIS (Infections and infestations) | 5
INJECTION SITE PAIN (General disorders) | 79
INJECTION SITE PRURITUS (General disorders) | 12
INJECTION SITE REACTION (General disorders) | 35
INJECTION SITE URTICARIA (General disorders) | 1
ALLERGIC REACTION (General disorders) | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 1
FEVER (General disorders) | 25
RIGORS (General disorders) | 2
MIGRAINE (Nervous system disorders) | 1
DYSPEPSIA (Gastrointestinal disorders) | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1
GASTROENTERITIS (Gastrointestinal disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 21
HERPES ZOSTER (Infections and infestations) | 1
PHARYNGITIS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
COUGHING (Respiratory, thoracic and mediastinal disorders) | 2
URTICARIA (Skin and subcutaneous tissue disorders) | 1
LEUCOPENIA (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.